CLINICAL TRIAL: NCT04823936
Title: Effect of Core Stability on Balance and Coordination on Ataxic Cerebral Palsied Children
Brief Title: Core Stability in Ataxic Cerebral Palsied Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ali, associate professor of physical therapy Faculty of Physical Therapy Cairo University, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Faculty of Physcial therapy
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Ataxic Cerebral Palsied Children; Core Stability; Balance and Coordination; Severity of the Ataxia
Keywords: Ataxia; humac balance sysytem; balance; coordination
MeSH Terms: conditions — Ataxia

STUDY DESIGN:
Intervention Model Description: pre-test post-test randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): received the selected physical therapy program for one hour, three times weekly for two successive months including facilitation of balance and protective reactions from kneeling, half kneeling and standing position, standing alone on balance board, standing on one leg, open gait training alone (walking on the balance beam, walking on the stepper and walking on wedges), training stair climbing, and strengthening of the back and abdominal muscles.
- study group (Active Comparator): received the selected physical therapy program for one hour, three times weekly in addition to core stability training program for 30 minutes
  Interventions: Other: core stability training

INTERVENTIONS:
Other: core stability training — core stability training program for 30 minutes including Supine abdominal draw in Abdominal draw in with double knee to chest Trunk twist while sitting on medical ball Lying supine on the medical ball and rotating the trunk to the sides Contracting abdominal muscles while lying in a supine position and pulling the limbs upward with arms and legs kept close Bringing up the arms and legs simultaneously in the prone position Bridging with head on medical ball hold this position for 3-5 s then slowly relaxes Bridging while shoulders and hands are on the floor and one leg is raised Lying supine on the medical ball and holding the abdomen in and bringing with one leg up
  Other Names: selected physical therapy program
  Arms: study group

SUMMARY:
Forty children with cerebellar ataxia ranged in age from five to nine years old, they were randomly assigned into two matched control and study groups. The control groups received the selected physical therapy program three times weekly one hour per session while the study group received core stability training for 30 minutes in addition to the selected physical therapy program. Both groups were evaluated by SARA Scale for the Assessment and Rating of Ataxia, Balance Error Scoring Systems scale, Bruininks-Oseretsky test of motor Proficiency 2ed subtest 4 (bilateral coordination), and subtest 7 (upper limb coordination), and HUMAC Balance System before and after two months of intervention.

DETAILED DESCRIPTION:
Forty ataxic cerebral palsied children were selected from private pediatric physical therapy centers, their ages ranged from five to nine years old. They were simply randomly assigned into two matched control and study group via an electronic program (SPSS) as illustrated in figure (1). The selected children had level IV according to the gross motor function classification system and their ataxia severity score was less than 25 according to the scale for the Assessment and Rating of Ataxia (SARA). Children have excluded it they had visual impairment, spasticity, uncontrolled convulsions, any other neuromuscular diseases, ataxia-telangiectasia, spinocerebellar ataxia, and Joubert syndrome.

Measures

1. Scale for the Assessment and Rating of Ataxia (SARA): it is a clinical scale that assesses a range of different impairments in cerebellar ataxia. The scale is made up of 8 items related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements, and heel-shin test [22].
2. Balance Error Scoring Systems scale (BESS): This tool assesses postural control in stable surfaces the tests performed on the ground and foam block. It composes of six items performed with eyes closed taking 20 Sc each [23].
3. The Bruininks-Oseretsky Test of Motor Proficiency 2ed (BOT-2): It is a standardized, norm-referenced measure used by physical therapists and occupational therapists in the clinic and school practice settings. It is an individually administered test that delivers a most precise measure of motor skills, both gross and fine, of children and youth, 4 through 21 years of age [24].
4. HUMAC Balance System: Developed by Computer Sports Medicine, Inc. (CSMi), The HUMAC Balance System is a high-quality computerized balance system. It is a static force plate (Force Plate Mode) that measures Center of Pressure (COP) and Force [25].

1- Procedures for evaluation Both groups were evaluated before and after two months of intervention by the SARA Scale for the Assessment and Rating of Ataxia, Balance Error Scoring Systems scale, Bruininks-Oseretsky test of motor Proficiency 2ed subtest 4 (bilateral coordination) and subtest 7 (upper limb coordination), and HUMAC Balance System.

2- Procedure for intervention The Control group received the selected physical therapy program for one hour, three times weekly for two successive months including facilitation of balance and protective reactions from kneeling, half kneeling and standing position, standing alone on balance board, standing on one leg, open gait training alone (walking on the balance beam, walking on the stepper and walking on wedges), training stair climbing, and strengthening of the back and abdominal muscles.

The study group received the selected physical therapy program for one hour, three times weekly in addition to core stability training program for 30 minutes [26]. The core stability training program.

illustration of core stability program. Supine abdominal draw in 10- 15 times Abdominal draw in with double knee to chest 10- 15 times Trunk twist while sitting on medical ball 10- 15 times Lying supine on the medical ball and rotating the trunk to the sides 10- 15 times Contracting abdominal muscles while lying in a supine position and pulling the limbs upward with arms and legs kept close 10- 15 times Bringing up the arms and legs simultaneously in the prone position 10- 15 times Bridging with head on medical ball hold this position for 3-5 s then slowly relaxes 10- 15 times Bridging while shoulders and hands are on the floor and one leg is raised 10- 15 times Lying supine on the medical ball and holding the abdomen in and bringing with one leg up 10- 15 times

ELIGIBILITY:
Inclusion Criteria:

* ataxic cerebral palsied children
* must have level IV according to the gross motor function classification system.

Exclusion Criteria:

* spastic cerebral palsied children
* ataxia-telangiectasia
* spinocerebellar ataxia
* Joubert syndrome.
* sensory ataxic

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — boys and girls ranged in age from five to nine years old
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
HUMAC Balance System | 2 months
  measuring Mobility Standing Balance Bilateral, stability standing balance bilateral, limit of stability and modified clinical test of sensory integration of balance Stabil
The Bruininks-Oseretsky Test of Motor Proficiency (bilateral coordination subtest) | 2 months
  measuring bilateral coordination with maximum score of the subtest 24 the higher scale score indicates better bilateral coordination
The Bruininks-Oseretsky Test of Motor Proficiency (upper limb coordination subtest) | 2 months
  measuring upper limb coordination with maximum score of the subtest 39 and higher sub test score indicate more upper limb coordination

SECONDARY OUTCOMES:
Balance Error Scoring Systems scale | 2 months
  measuring balance with maximum score of the scale 60 the higher scale score indicated more balance loss and increased severity of the cases.
Scale for the Assessment and Rating of Ataxia | 2 months
  measuring severity of ataxia with maximum score of the scale 40 the higher score of the scale means sever affected ataxic child

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No